CLINICAL TRIAL: NCT03369431
Title: The Efficacy of the Multistrain Probiotic, Vivomixx, on Behaviour and Gastrointestinal Symptoms in Children With Autism Spectrum Disorder (ASD)
Brief Title: Efficacy of Vivomixx on Behaviour and Gut Function in Autism Spectrum Disorder
Acronym: VIVO-ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17/0148
Record Dates: First submitted 2017-11-27; First posted 2017-12-12 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Gastrointestinal; behaviour; constipation; diarrhoea; probiotic; sociability
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Behavior; Constipation; Diarrhea

STUDY DESIGN:
Intervention Model Description: 3-month randomised controlled cross-over design with 4-week washout. Outcomes measured at baseline and last week of each treatment phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vivomixx, then placebo (Other): This group starts with Vivomixx probiotic for the first 12 weeks then crosses over to have the placebo after a 4-week washout.
  Interventions: Dietary Supplement: Vivomixx; Dietary Supplement: Placebo
- Placebo, then Vivomixx (Other): This group starts with the placebo for the first 12 weeks then crosses over to have Vivomixx probiotic after a 4-week washout.
  Interventions: Dietary Supplement: Vivomixx; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx — Multi-strain probiotic containing 450 billion lyophilized bacterial cells per sachet belonging to 8 probiotic strains. The probiotic strains contained in the intervention are Streptococcus thermophilus, Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasei, Lactobacillus delbrueckii subsp. bulgaricus.
Dietary Supplement: Placebo — 4.4 grams of maltose and silicon dioxide per sachet

SUMMARY:
The purpose of this study is to assess the effects of 3 months supplementation with the multi strain probiotic Vivomixx on the overall function, aberrant behaviours and frequency of gastrointestinal symptoms in children with Autism Spectrum Disorders and co-morbid gastrointestinal symptoms.

The investigators will also assess the effect of the intervention on parenting stress.

A further issue will be to identify any predictors of response to the probiotic.

Finally, the investigators will assess whether there is an association between altered behaviour and altered gut function in users of Vivomixx.

DETAILED DESCRIPTION:
Potential trial participants will be recruited via one of two routes,

1. A children's charity will email parents of children with ASD on their database with a copy of our recruitment poster and asked to contact us if they wish their child to be considered for the study.
2. Information on the trial was given to attendees of a bi-annual charity conference in June 2016 run by Thinking Autism charity, which offers support to parents of children with ASD. Contact details were taken from parents who were potentially interested in their child taking part. They will be emailed a copy of the recruitment poster and asked to contact the investigators if they wish their child to be considered for the study.

Parents who respond to the recruitment poster will be emailed the Patient Information Sheet and the Child Information Leaflet. A few days later, they will then be emailed to ask if they are interested in answering some questions to see if their child is eligible for the study. If they are, an appointment will be made to phone them and complete the screening questionnaire. For those children that fit the requirements for the trial, the parents will be invited for their child to take part. The participants recruited to the study will be allocated at random to either group A or B and will be given a unique Study Number. All data collected throughout the study will be anonymised and identified only by the participant's study number.

The first week of study will be a taste evaluation of the product for all participants (both groups). The taste evaluation is to ensure that the participant finds the taste acceptable and is willing to take the treatment product. For those that find the taste acceptable they will then either receive a 12-week course of Vivomixx probiotic or a 12-week course of the placebo powder, according to their random group allocation. The placebo powder has the same look and taste as Vivomixx.

Once the participant has passed the taste evaluation, the child's educator will be sent a letter inviting them to participate in the study. Included with this letter will be a consent slip, a copy of the Educator Questionnaire and a stamped addressed envelope for returning the questionnaires and consent slip to the researcher.

All participants' parents will be phoned by the researcher in Weeks 5 and 9 to adjust the treatment dose, offer support and check compliance.

Those parents whose child is eligible but who choose not to take part will be asked for the main reason and this will be logged in the screening log of patients.

After 12 weeks there will be 4 weeks when neither group is taking any treatment (a washout period). After this, participants who complete all 12 weeks of the double-blind treatment period will be eligible to enter the double-blind 12-week withdrawal period. The participants that have been taking the placebo will then receive a 12-week course of Vivomixx probiotic. The participants that have received Vivomixx, will take a 12-week course of the placebo. All participants' parents will be phoned by the researcher in Weeks 21 and 25 to adjust the treatment dose, offer support and check compliance. We will also ask about their experience of the study.

The investigators are primarily interested in whether participants in the intervention group (Vivomixx) have had more of an improvement in their overall function after their 12-week course of Vivomixx compared to that of the control group (receiving the placebo). The investigators will also measure the effect of the active treatment on parent stress compared to the control group and the effect of the active treatment on gastrointestinal symptoms and clinician's global assessment compared to the control group.

During the study the investigators will assess how well the participants kept to the treatment plan. The investigators will also record changes that happen during the trial that may affect the efficacy of treatment, for example taking antibiotics or a significant change in diet. The investigators will talk to the participant's parents to find how they perceived the treatment and how their child tolerated the treatment.

Statistical methodology and analysis The intention-to-treat (ITT) analysis will be performed on all participants who are randomised. An additional analysis will be done on only those participants who complete the study per protocol analysis. Details of the statistical analysis is given in the Statistical Analysis Plan.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of ASD confirmed by a medical professional using one of the following standard assessment tools: Autism Diagnostic Interview - Revised (ADI-R), Diagnostic Interview for Social and Communication disorders (DISCO), Developmental, Dimensional and Diagnostic Interview (3di) or Autism Diagnostic Observation Schedule (ADOS).
* Have one or more gastrointestinal symptoms (constipation, diarrhoea, abnormal stools, pain on defecation, abdominal pain, gaseousness/bloating, reflux) for the past 6 months.
* Are either not taking any medication or have been on the same medication for the last 3 months.
* The patient or the patient's parents/guardian are willing and able to provide a written informed consent
* Be willing and able to continue with current medication or nutritional supplements throughout the 30-week trial.
* The patient's primary carer must be willing and able to complete the questionnaires at three time-points in the study. These questionnaires are only available in written English.
* Be willing to refrain from starting any kind of special diet for the duration of the study.
* Be between 3 years and 16 years of age

Exclusion Criteria:

* Has a diagnosis of Retts Syndrome or Fragile X
* Aged over 16 years or under 3 years
* On NSAIDs
* Taken antibiotics in the past month
* Taken a probiotic in the past month
* History of intolerance or allergy to probiotics
* The patient's primary carer is not willing or are not able to complete the questionnaires at three time-points in the study. These questionnaires are only available in written English.
* Has taken part in a clinical trial in the past 3 months

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton V Emmanuel, MBBS, FRCP, Principal Investigator — University College, London
Locations (1):
- University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vivomixx, Then Placebo | Placebo, Then Vivomixx
Started | 35 | 34
Taste Test (1 Week) | 35 | 34
Part 1 Treatment (12 Weeks) | 34 | 34
Washout (4 Weeks) | 34 | 32
Part 2 Treatment (12 Weeks) | 34 | 32
Completed | 31 | 27
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vivomixx, Then Placebo | Placebo, Then Vivomixx | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean age | 8.3 (2.3) | 7.3 (2.9) | 7.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 31 | 26 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic origin: Arab | 1 | 1 | 2
  Ethnic origin: Asian/Asian British | 3 | 3 | 6
  Ethnic origin: Black/African/Caribbean/Black British | 2 | 2 | 4
  Ethnic origin: Chinese | 0 | 1 | 1
  Ethnic origin: Hispanic | 0 | 1 | 1
  Ethnic origin: Mixed/Multiple ethnic | 8 | 4 | 12
  Ethnic origin: White | 21 | 22 | 43
Autism Treatment Evaluation Checklist Total score [Mean (Standard Deviation); unit: score on a scale] — The Autism Treatment Evaluation Checklist (ATEC) total score is a measure of global function. The Total score ranges from 0-180. A lower score indicates a greater level of global function. The four sub scales of the ATEC are summed to calculate the Total score.
  score on a scale | 70.15 (25.28) | 76.32 (30.18) | 73.24 (27.80)

OUTCOME MEASURES:

1. Primary Outcome: A Change in the Autism Treatment Evaluation Checklist (ATEC) Total Score Compared to Baseline.
Description: The ATEC is a one-page form, designed to be completed by parents, teachers, or caregivers. It consists of 4 subtests: I. Speech/Language Communication (14 items); II. Sociability (20 items); III. Sensory/ Cognitive Awareness (18 items); and IV. Health/Physical/Behavior (25 items). The scale covers 77 items and gives a total score and scores for each of the 4 sub-sections. The higher the score, the greater the impairment overall or in a sub-section. The ATEC total score can range from 0 - 180 and is calculated by summing the scores of each subsection.
Time Frame: ATEC will be measured at the time of enrolment to the study, after the first 12-week treatment and after the second 12-week treatment by the child's primary carer and also by the child's educator.
Population: All participants who received at least one dose of each intervention and whose primary carer at least completed the ATEC questionnaire at enrolment and after Part 1 treatment. Those who were withdrawn or lost-to-followup in Part 2 (n=6) were assumed to have no change from their last ATEC score.
Measure: Mean (Standard Deviation); unit: percentage change from baseline score
Groups:
- Vivomixx: Participants who received Vivomixx at an age-group determined dose.
- Placebo: Participants who received Placebo powder at an age-group determined dose
Arm/Group | Vivomixx | Placebo
Number analyzed (Participants) | 64 | 64
percentage change from baseline score | -12.122 (20.9140) | -11.427 (20.3055)
Statistical Analysis 1: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the percentage change from baseline in the ATEC Total between Vivomixx and Placebo. A sample size of 72 participants was needed to determine an effect size of 0.50 with 80% power, with a type 1 error of 5% using a two-sided test. This calculation is based on the assumed effect size of the primary outcome measure, the ATEC. The minimally clinically important difference based on the primary outcome measure with this instrument was 15 points; Test type: Superiority; p = 0.784, t-test, 2 sided

2. Secondary Outcome: The Change in the Frequency of Gastrointestinal Symptoms Compared to Baseline, as Measured by the Gastrointestinal History (GIH) Questionnaire.
Description: In 2003 the Childhood Autism Risks from Genetics and the Environment (CHARGE) study developed and began using a frequency assessment of GI symptoms in autistic children, which they called the Gastrointestinal History Questionnaire. The Gastrointestinal History questionnaire (GIH) includes 10 Likert scale items for the following symptoms: abdominal pain, gaseousness/bloating sensation, diarrhoea, constipation, pain on stooling, vomiting, difficulty swallowing, blood in stools and blood in vomit. These have been equated to a numerical score as follows; never=0, rarely=1, sometimes=2, frequently=3, always=4.
Time Frame: GIH will be measured at the time of enrolment to the study, after the first 12-week treatment and after the second 12-week treatment.
Population: All participants who received at least one dose of each intervention and whose primary carer completed at least a GIH at enrolment and after Part 1 treatment. Those who were withdrawn or lost-to-followup in Part 2 (n=6) were assumed to have no change since their last GIH was completed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vivomixx | Placebo
Number analyzed (Participants) | 66 | 66
units on a scale
  Change in abdominal pain frequency | -0.92 (0.128) | -0.82 (0.128)
  Change in gaseousness frequency | -0.70 (0.159) | -0.86 (0.157)
  Change in diarrhoea frequency | -0.92 (0.149) | -0.80 (0.153)
  Change in constipation frequency | -0.92 (0.176) | -1.00 (0.153)
  Change in pain on stooling frequency | -0.92 (0.158) | -0.82 (0.160)
  Change in difficulty swallowing frequency | -0.12 (0.063) | -0.08 (0.084)
  Change in vomiting frequency | -0.27 (0.095) | -0.23 (0.094)
  Change in blood in stool frequency | -0.06 (0.048) | -0.06 (0.043)
  Change in blood in vomit frequency | -0.02 (0.015) | -0.02 (0.015)
Statistical Analysis 1: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline in frequency of Abdominal Pain between Vivomixx and Placebo; Test type: Superiority; p = 0.357, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 2: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline in frequency of Gaseousness between Vivomixx and Placebo; Test type: Superiority; p = 0.290, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 3: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline in frequency of Diarrhoea between Vivomixx and Placebo; Test type: Superiority; p = 0.418, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 4: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline in frequency of Constipation between Vivomixx and Placebo; Test type: Superiority; p = 0.734, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 5: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline in frequency of Pain on Stooling between Vivomixx and Placebo; Test type: Superiority; p = 0.362, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 6: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline in frequency of Difficulty Swallowing between Vivomixx and Placebo; Test type: Superiority; p = 0.705, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 7: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in change from baseline in frequency of vomiting between Vivomixx and placebo; Test type: Superiority; p = 0.589, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 8: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in change from baseline in frequency of blood in stool between Vivomixx and placebo; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon signed rank
Statistical Analysis 9: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in change from baseline in frequency of blood in vomit between Vivomixx and placebo; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon signed rank

3. Secondary Outcome: A Change in the Aberrant Behaviour Checklist (ABC) Section Scores Compared to Baseline.
Description: Maladaptive behavior will be measured using five subscales of the ABC: Irritability (15 items), Lethargy/social withdrawal (16 items), Stereotypic behaviour (7 items), Hyperactivity/Noncompliance (16 items) and Inappropriate speech (4 items). A higher score indicates greater difficulty. The minimum score for each section is 0. The maximum scores for the sections are: Irritability 45, Lethargy/social withdrawal 48, Stereotypic behaviour 21, Hyperactivity/Noncompliance 48 and Inappropriate speech 12.
Time Frame: ABC was measured at the time of enrolment to the study, after the first 12-week treatment and after the second 12-week treatment by the child's primary carer.
Population: All participants who received at least one dose of each intervention and whose primary carer at least completed the ABC questionnaire at enrolment and after the Part 1 treatment. Those who were withdrawn or lost-to-follow-up in Part 2 were assumed to have no change from their last ABC questionnaire.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vivomixx | Placebo
Number analyzed (Participants) | 62 | 62
score on a scale
  Change in Irritability | -3.00 (1.100) | -3.05 (1.065)
  Change in Lethargy/social withdrawal | -2.26 (0.842) | -3.11 (.780)
  Change in stereotypic behaviour | -1.06 (0.404) | -1.08 (0.399)
  Change in Hyperactivity/Noncompliance | -2.42 (0.944) | -2.16 (0.894)
  Change in Inappropriate speech | -0.45 (0.290) | -0.37 (0.316)
Statistical Analysis 1: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline of ABC Irritability score between Vivomixx and Placebo; Test type: Superiority; p = 0.635, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 2: Comparison: Vivomixx vs Placebo; The null hypothesis is that there is no difference in the change from baseline of ABC Lethargy/social withdrawal score between Vivomixx and Placebo; Test type: Superiority; p = 0.367, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 3: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline in the ABC Stereotypic behaviour between Vivomixx and Placebo; Test type: Superiority; p = 0.609, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank
Statistical Analysis 4: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline of the ABC Hyperactivity/Noncompliance between Vivomixx and Placebo; Test type: Superiority; p = 0.805, t-test, 2 sided; Paired samples t-test
Statistical Analysis 5: Comparison: Vivomixx vs Placebo; Null hypothesis is that there is no difference in the change from baseline of the ABC Inappropriate Speech between Vivomixx and Placebo; Test type: Superiority; p = 0.985, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank test used

4. Secondary Outcome: The Change in the Autism Parenting Stress Index (APSI) Score Compared to Baseline.
Description: This one-page, self-assessment questionnaire was developed and validated in 2012. It is designed to assess parent stress in 13 aspects of autism of concern to parents and to provide a measure of parenting stress specific to core symptoms of autism and common co-occurring issues. It reflects the time, effort and actual difficulty of parenting in the light of the physical, social and communication barriers imposed by autism. It is intended for use by clinicians to assess the effects of an intervention on parenting stress. A higher score indicates greater parenting stress. The minimum score is 0 and the maximum score is 65.
Time Frame: APSI will be measured at the time of enrolment to the study, after the first 12-week treatment and after the second 12-week treatment.
Population: All participants who received at least one dose of each intervention and whose primary carer at least completed the APSI at enrolment and after Part 1 treatment. Those who were withdrawn or lost-to-followup in Part 2 were assumed to have no change since their last APSI was completed.
Measure: Mean (Standard Error); unit: difference in score on a scale from base
Arm/Group | Vivomixx | Placebo
Number analyzed (Participants) | 64 | 64
difference in score on a scale from base | -3.73 (0.928) | -3.11 (0.872)
Statistical Analysis 1: Comparison: Vivomixx vs Placebo; Test type: Superiority; p = 0.661, Wilcoxon (Mann-Whitney); Related-samples Wilcoxon Signed Rank

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vivomixx | Placebo
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/68
Other Adverse Events (participants affected / at risk) | 10/66 | 16/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivomixx (N=66) | Placebo (N=68)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (5)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Worsening behaviour (General disorders) | 2 (2) | 3 (3)
Temporary poor sleep (General disorders) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 2 (2) | 3 (3)
Loose stools (Gastrointestinal disorders) | 3 (3) | 1 (1)
Food intolerance reaction (Immune system disorders) | 0 (0) | 1 (1)
Persistent cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Increased sensory sensitivity (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Too few ATEC and ABC questionnaires were completed by educators to enable analysis.

Stool sample collection was disrupted by Covid-19 lockdown and consequently there were insufficient samples for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT03369431/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT03369431/SAP_001.pdf